CLINICAL TRIAL: NCT01141517
Title: Predictors of Smoking Cessation Among Teen Smokers
Brief Title: Predictors of Teen Smoking-cessation
Acronym: NOT
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Brady Reynolds, Associate Professor, University of Kentucky
Other Study IDs: IRB09-00538; 5R01DA023087-02 (NIH)
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cigarette Smoking
Keywords: adolescent quit-smoking program.
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Not-On-Tobacco smoking cessation program — Adolescent quit-smoking program; Not-On-Tobacco

SUMMARY:
The primary objective of this research is to explore relations between impulsive behavior and smoking-cessation success among treatment-seeking teens enrolled in a quit-smoking program.

It is hypothesized that teens who do not successfully stop smoking (or who drop out of the treatment program) will be more impulsive (from measures taken just prior to treatment) than those who do successfully stop or significantly reduce rate of smoking.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 13 and 19
* Enrolled in the NOT program offered by Nationwide Children's Hospital
* Currently smoke at least one cigarette per day

Exclusion Criteria:

* Adolescents must be English speaking

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will be adolescent smokers between the ages of 13-19 recruited from local high-schools (Franklin county; Pike county, and Scioto County in Ohio), shopping malls, and newspaper ads.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of adolescents that quit/reduce smoking and those who do not quit/reduce. | 8.5 months
  Primary outcomes will be the number of adolescents who quit or reduced smoking and the number of adolescents who did not quit or reduce.

CONTACTS AND LOCATIONS:
Overall Officials: Brady A Reynolds, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States